CLINICAL TRIAL: NCT07248865
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose (SAD) and Multiple-Ascending-Dose (MAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Injection(s) of CLYM116 in Normal Healthy Volunteers
Brief Title: A Phase 1 Study of CLYM116 in Normal Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Climb Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CLYM116-NHV-101
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
Keywords: CLYM116; APRIL; monoclonal antibody; healthy volunteers; Phase 1; IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CLYM116 (Experimental): Subcutaneous (SC) injection of CLYM116
  Interventions: Drug: CLYM116
- Placebo (Placebo Comparator): Subcutaneous (SC) injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CLYM116 — CLYM116 to be administered by SC injection
  Arms: CLYM116
Drug: Placebo — Placebo solution to be administered at a matching volume by SC injection
  Arms: Placebo

SUMMARY:
This Phase 1, first-in-human study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of CLYM116 in healthy volunteers.

DETAILED DESCRIPTION:
CLYM116 is a humanized monoclonal antibody that selectively binds to a proliferation inducing ligand (APRIL). This is a Phase 1, randomized, double-blind, placebo-controlled, single-center study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of CLYM116 in adult normal healthy volunteers (NHVs). The study will enroll up to 48 subjects, across up to five cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females aged 18-60 years, inclusive
* Body mass index (BMI) between 18 and 32 kg/m² and weight between 45 and 110 kg
* Clinically normal medical history, physical exam, ECG, and laboratory results (or abnormalities deemed not clinically significant)
* Willing and able to comply with study procedures and provide informed consent
* Women of childbearing potential must use highly effective contraception and have negative pregnancy tests
* Men must use contraception and refrain from sperm donation for 4 months post-dose
* Completion of COVID-19 vaccination according to local guidelines, as well as influenza vaccination (within 12 months)

Exclusion Criteria:

* Prior treatment with investigational drugs within 30 days or 5 half-lives
* Previous or current hypogammaglobulinemia
* Current presence of allergic reactions considered clinically significant
* Positive tests for HIV, hepatitis B/C, syphilis, or tuberculosis
* Tobacco use (>2 cigarettes/day), alcohol abuse, or drug abuse
* Recent live vaccination (within 21 days) or any non-live vaccine (within 14 days)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple ascending doses of CLYM116 in healthy volunteers Incidence of treatment-emergent adverse events | From Screening through to Day 85, or final follow-up visit
Incidence of injection site reactions Number of injection site reactions | From Baseline through to Day 4 and Day 15 to Day 18

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) Measurement of the maximum observed plasma concentration. | From Baseline through to Day 85 (except Day 14), or final follow-up visit
Time to Maximum Observed Concentration (Tmax) Measurement of the time to maximum observed concentration. | From Baseline through to Day 85 (except Day 14), or final follow-up visit
Area Under the Curve (AUC) Measurement of the area under the drug concentration-time curve. | From Baseline through to Day 85 (except Day 14), or final follow-up visit.
Half-Life (T1/2) Measurement of the half-life in days | From Baseline through to Day 85 (except Day 14), or final follow-up visit
Levels of Immunoglobulins Measurement of Immunoglobulins and changes over time | From Screening through to Day 85, or final follow-up visit
Level of APRIL Measurement of APRIL in pg/mL and changes over time | Day -1, Baseline, Day 1, Day 4, Day 8, Day 14, Day 15, Day 17, Day 18, Day 22, Day 29, Day 71, day 85, final follow up visit
Immunogenicity Measurement of CLYM116 antidrug antibodies (ADA) | Baseline, Day 15, Day 29, Day 43, Day 71, Day 85, follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Brisbane, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No